CLINICAL TRIAL: NCT02096783
Title: Randomized-Controlled, Pilot Study of the Effects of a Brief, Scripted Sexual Health Intervention on Sexual Function for Women With Gynecologic Cancer
Brief Title: Scripted Sexual Health Informational Intervention in Improving Sexual Function in Patients With Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW13080; NCI-2014-00471 (Registry Identifier: NCI Trial ID); UW13080 (Other: University of Wisconsin Carbone Cancer Center); P30CA014520 (NIH); 2014-0122 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL/OBSTET (Other: UW Madison)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-11

CONDITIONS: Anxiety Disorder; Cervical Cancer; Endometrial Cancer; Female Reproductive Cancer; Gestational Trophoblastic Tumor; Ovarian Epithelial Cancer; Ovarian Germ Cell Tumor; Sexual Dysfunction; Uterine Sarcoma; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Anxiety Disorders; Uterine Cervical Neoplasms; Endometrial Neoplasms; Gestational Trophoblastic Disease; Carcinoma, Ovarian Epithelial; Sexual Dysfunction, Physiological; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (standard counseling) (Active Comparator): Patients receive standard counseling at both the pre-operative and 2-4 week post-operative visit.
  Interventions: Other: counseling intervention; Other: questionnaire administration
- Arm II (standard counseling, scripted intervention) (Experimental): Patients receive standard counseling at the pre-operative visit and the scripted sexual health intervention at the 2-4 week post-operative visit.
  Interventions: Other: informational intervention; Other: counseling intervention; Other: questionnaire administration
- Arm III (standard counseling, scripted intervention) (Experimental): Patients receive standard counseling and the scripted sexual health intervention at the pre-operative visit and standard counseling at the 2-4 week post-operative visit.
  Interventions: Other: informational intervention; Other: counseling intervention; Other: questionnaire administration
- Arm IV (standard counseling, scripted intervention) (Experimental): Patients receive standard counseling and the scripted sexual health intervention at both the pre-operative and 2-4 week post-operative visit.
  Interventions: Other: informational intervention; Other: counseling intervention; Other: questionnaire administration

INTERVENTIONS:
Other: informational intervention — Given scripted intervention
  Arms: Arm II (standard counseling, scripted intervention); Arm III (standard counseling, scripted intervention); Arm IV (standard counseling, scripted intervention)
Other: counseling intervention — Given standard counseling
  Other Names: counseling and communications studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the feasibility of a pre-operative and/or post-operative scripted sexual health informational intervention and how well it works in improving sexual function in patients with gynecologic cancer. Discussing sexual outcomes and counseling options with patients may help improve sexual outcomes and/or anxiety after primary gynecologic cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of patient recruitment, including time required to consent, enroll and retain the necessary number of participants.

II. To determine the distribution of candidate primary patient-reported outcome measures, including time to resumption of sexual activity, global satisfaction with sex life, sexual function and anxiety in this particular population.

III. To establish the prevalence of patient recall of the intervention to determine the most effective time at which to deliver the intervention.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive standard counseling at both the pre-operative and 2-4 week post-operative visit.

ARM II: Patients receive standard counseling at the pre-operative visit and the scripted sexual health intervention at the 2-4 week post-operative visit.

ARM III: Patients receive standard counseling and the scripted sexual health intervention at the pre-operative visit and standard counseling at the 2-4 week post-operative visit.

ARM IV: Patients receive standard counseling and the scripted sexual health intervention at both the pre-operative and 2-4 week post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new suspected or confirmed gynecologic malignancies
* Patients plan to have primary surgery at either the University of Chicago Hospital or the University of Wisconsin Hospital
* Patients must be English speaking

Exclusion Criteria:

* Previous treatment of any cancer excluding skin cancer
* Patients with a suspected benign gynecologic process
* Patients who are prisoners or incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of patient recruitment | Up to 9 months
  To inform possible issues in recruitment for a large-scale randomized controlled trial, the ratio of enrolled subjects to total eligible potential subjects as well as the time necessary to recruit those subjects will be tracked.

SECONDARY OUTCOMES:
Resumption of sexual activity after cancer surgery | Up to 9 months
  Resumption of sexual activity after cancer surgery will be measured using items adapted from a previous national, multi-site study of sexual outcomes following an acute myocardial infarction.
Retention | Up to 9 months
  The percentage of subjects completing the final assessment from the total number of subjects enrolled will be calculated.
Satisfaction with sex life independent of specific sexual function measured by Patient Reported Outcomes Measurement Information System (PROMIS) Global Satisfaction with Sex Life questionnaire | Up to 9 months
  Descriptive statistics will be used to summarize survey responses overall and separately for both the experimental and control arms.
PROMIS Sexual Function Profile | Up to 9 months
  Descriptive statistics will be used to summarize survey responses overall and separately for both the experimental and control arms.
Recall of intervention | Up to 9 months
  Subjects will be queried to learn whether they recall receiving physician counseling about sexual health outcomes after surgery with follow up questions regarding whether or not the patient has spoken with other healthcare providers about sexual concerns.
Patient-reported anxiety measured by PROMIS Anxiety 4a short form | Up to 6 months
  Descriptive statistics will be used to summarize survey responses overall and separately for both the experimental and control arms.
Rate of referral acceptance | Up to 9 months
  The rate of acceptance of sexual health clinic referrals as well as rates of utilization of these referrals will be tracked using medical record abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: David Kushner, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/